CLINICAL TRIAL: NCT02412644
Title: Efficacy and Safety of Combining Apremilast 30mg Bid With Narrowband UVB in the Treatment of Moderate-to-severe Plaque Psoriasis
Brief Title: Apremilast 30mg Bid With Narrowband UVB in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-CL-PSOR-PI-004893
Record Dates: First submitted 2015-02-23; First posted 2015-04-09 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-12

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apremilast + apremilast (Active Comparator): apremilast 30mg bid for 12 weeks.followed by apremilast 30 mg bid for 24 weeks
  Interventions: Drug: apremilast
- apremilast + placebo (Placebo Comparator): apremilast 30mg bid for 12 weeks followed by placebo bid for 24 weeks
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast

SUMMARY:
12 weeks open label with Otezla® and NUVB, followed by 6 month double blind Otezla® (apremilast) or placebo to subjects who obtain PASI 75 at week 12 of phototherapy

DETAILED DESCRIPTION:
Primary Objective: To evaluate the effectiveness of Otezla (apremilast®) in promoting maintenance of response in those subjects who obtained PASI-75 at week 12 of phototherapy.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet the following criteria to be enrolled in this study:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of chronic plaque-type
3. Moderate to severe plaque type psoriasis as defined at baseline by:

   * PASI score of 12 or greater,
   * PGA score of 3 or greater
   * BSA affected by plaque-type psoriasis of 10% or greater,
4. Able and willing to give written informed consent prior to performance of any study-related procedures

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in this study:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic, and/or guttate psoriasis) or drug induced psoriasis
2. Subjects with previous exposure to apremilast
3. Malignancy or history of malignancy, except for:

   * treated [ie, cured] basal cell or squamous cell in situ skin carcinomas;
   * treated [ie, cured] malignancy with no evidence of recurrence within the previous 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, MD, Principal Investigator — Psoriasis Treatment Center of Central New Jersey
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment May 28 2015-November 2015 through practice database
Groups:
- Apremilast + Apremilast: apremilast 30 mg BID for 12 weeks + apremilast 30 mg BID through week 36
- Apremilast + Placebo: apremilast 30 mg BID for 12 weeks + placebo BID through week 36
Period: Overall Study
Arm/Group | Apremilast + Apremilast | Apremilast + Placebo
Started | 21 | 8
Completed | 6 | 4
Not Completed | 15 | 4

BASELINE CHARACTERISTICS:
Groups:
- Apremilast + Apremilast: apremilast + apremilast 30mg bid after week 12
- Apremilast + Placebo: apremilast + Placebo bid after week 12
- Total: Total of all reporting groups
Arm/Group | Apremilast + Apremilast | Apremilast + Placebo | Total
Number analyzed (Participants) | 21 | 8 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (22) | 55 (38) | 47 (50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 12 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 6 | 21
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 21 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Maintaining Psoriasis Area Severity Index Score (PASI) 75 at Week 36
Description: Analysis of Psoriasis Area Severity Index Score at week 36 to determine number of subjects who maintained PASI 75 at week 36
Time Frame: 36weeks
Measure: Number; unit: participants
Groups:
- Apremilast + Apremilast: apremilast + apremilast
- Apremilast + Placebo: apremilast + placebo
Arm/Group | Apremilast + Apremilast | Apremilast + Placebo
Number analyzed (Participants) | 6 | 4
participants | 4 | 2

2. Secondary Outcome: Number of Subjects Achieving Psoriasis Area Severity Index Score (PASI) 75 Response at Week 12
Description: Psoriasis Area Severity Score of 75 or greater at week 12
Time Frame: 12WEEKS
Population: 22 subjects completed week 12
Measure: Number; unit: participants
Groups:
- Apremilast: apremilast
Arm/Group | Apremilast
Number analyzed (Participants) | 22
participants | 16

3. Secondary Outcome: Number of Subjects Achieving Psoriasis Area Severity Index Score 90 at Week 36
Description: PASI 90 or greater at week 36
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | Apremilast + Apremilast | Apremilast + Placebo
Number analyzed (Participants) | 6 | 4
participants | 1 | 0

4. Secondary Outcome: Number of Subjects Achieving Physician Global Assessment Score of 0 or 1 at Week 36
Description: PGA score 0 or 1
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | Apremilast + Apremilast | Apremilast + Placebo
Number analyzed (Participants) | 6 | 4
participants | 1 | 0

ADVERSE EVENTS:
Groups:
- Apremilast 30mg BID First 12 Weeks: apremilast 30mg bid for 12 weeks
- Apremilast 30mg BID After 12 Weeks: apremilast bid after week 12
- Placebo BID After 12 Weeks: placebo bid after week 12
Arm/Group | Apremilast 30mg BID First 12 Weeks | Apremilast 30mg BID After 12 Weeks | Placebo BID After 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 13/29 | 3/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast 30mg BID First 12 Weeks (N=29) | Apremilast 30mg BID After 12 Weeks (N=8) | Placebo BID After 12 Weeks (N=8)
second degree burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — burn related NBUVB
Arterial rupture right leg (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — arterial rupture during catheterization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast 30mg BID First 12 Weeks (N=29) | Apremilast 30mg BID After 12 Weeks (N=8) | Placebo BID After 12 Weeks (N=8)
worsening of psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
First degree burn (Skin and subcutaneous tissue disorders) | 11 (19) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No